CLINICAL TRIAL: NCT02441270
Title: Evaluation of the Immunological Effects of a Combined Treatment With Radiation and Cyclophosphamide in Metastasized Breast Cancer Patients
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study was never started.
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC 2015/0204
Record Dates: First submitted 2015-04-24; First posted 2015-05-12 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Radiotherapy; Immunology
MeSH Terms: interventions — Cyclophosphamide; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide (Experimental)
  Interventions: Drug: Cyclophosphamide; Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Drug: Cyclophosphamide
Radiation: Stereotactic body radiotherapy

SUMMARY:
In metastasized of locally advanced breast cancer patients, local problems often occur like skin metastases, ulcerations or lymph node metastases. These problems are related to a worse quality of life, while overall survival is generally in the order of months to years. Treatment of these lesions is challenging, especially after failure of first or second line systemic therapy. Local treatments, like radiation, are able to give short-term palliation, but the effect is often disappointing in the long run. Therefore, the search for new therapeutic strategies like the combination of local and systemic treatments is emerging.

Recent investigations clearly show that radiation is capable of inducing a systemic anti-tumor response. Both in mouse models and in patients, it was reported that irradiating one metastasis can slow down the growth of other non-irradiated metastases. This effect is called the "abscopal effect" and is immune-mediated. There are also several chemotherapeutics that are capable of influencing the immune response like cyclophosphamide. Cyclophosphamide is a known inducer of immunogenic cell death, which leads to the activation of dendritic cells and thus the presentation of antigens.

In this pilot study the investigators wish to identify the immunological effects of combined treatment with radiation and cyclophosphamide in breast cancer patients. Five patients with metastasized breast carcinoma will be treated with the combined treatment and the immunological effects will be monitored using repeat blood draws and biopsies. These effects will be correlated to the clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of breast cancer
* Evidence of metastasized disease on imaging or during clinical examination
* Progressive disease during last systemic treatment
* Multiple (≥2) measurable lesions accessible for repeat biopsy, in particular:
* Skin- or subcutaneous metastases
* Lymph node metastases cervical, supraclavicular, axillary or inguinal
* Superficial lesions in the breast or on the thoracic wall
* Age ≥ 18 years
* Adequate organ and bone marrow function:
* ANC > 1500/µL
* haemoglobin > 9 g/dL (potentially after transfusion)
* thrombocytes ≥ 100 000/µL
* total bilirubin ≤ 1.5 X maximum reference value
* AST ≤ 2.5 X maximum reference value
* ALT ≤ 2.5 X maximum reference value
* creatinin ≤ 1.5 X maximum reference value
* Informed consent
* Chemotherapy or targeted therapy should be stopped for at least 1 month before the start of cyclophosphamide. Hormone therapy can be continued if it was not changed in the last 3 months

Exclusion Criteria:

* Life expectancy of less than 3 months or Karnofsky performance status < 70
* New line of systemic therapy planned
* Concomitant treatment with other experimental drugs
* Local therapies (radiation, surgery, topical anti-cancer treatment, intralesional therapy, laser treatment) at the target lesion(s) less than 4 weeks before the start of cyclophosphamide. Biopsy is allowed.
* Chemotherapy or targeted therapy < 4 weeks before the start of cyclophosphamide
* Hormone therapy change within the last 3 months
* Uncontrolled coagulation disorders
* Patients receiving therapeutic anticoagulants that cannot be stopped temporarily for repeat biopsy. Aspirin or anti-aggregants are allowed.
* Patients with a known immune-deficiency disorder or receiving immune-suppressive treatment
* Known allergy or intolerance for cyclophosphamide
* Pregnant or breastfeeding
* Women in the reproductive age not using a medically accepted method of contraception
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* Patient unlikely to comply with the protocol; i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Identification of the immunological effects, in peripheral blood and tumor biopsies, of the combined treatment with radiation and cyclophosphamide | 1.5 years
  Biopsies will be divided for 1) flowcytometric analysis (CD4 and CD8 tumor infiltrating lymphocytes, Tregs, dendritic cell subsets) and 2) immune histochemistry (CD8 tumor infiltrating lymphocytes, Foxp3+ Tregs).
  Immunomonitoring in peripheral blood by flow-cytometric analysis of leukocyte subsets involved in tumor-related immune responses: NK and T-cell subsets, dendritic cell subsets and myeloid-derived suppressor cells. Cytokine secretion patterns will be investigated using FACS and ELISA.
  Immune monitoring:
  Before the first session of radiation, 4 weeks after radiotherapy and 3 months after radiotherapy.

SECONDARY OUTCOMES:
Evaluation of the clinical/radiographical response of irradiated metastases | 1.5 years
  Evaluation of the clinical response of irradiated metastases will be done by monthly photographic documentation of all skin lesions.
  Evaluation of the radiographical response of irradiated metastases by 3-monthly imaging.
Evaluation of the response of non-irradiated metastases (the so-called "abscopal effect"). | 1.5 years
  Evaluation of the "abscopal effect" will be done by using the RECIST criteria and the immune related response criteria (irRC) 3 months post-radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital - Radiotherapy Department, Ghent, Belgium